CLINICAL TRIAL: NCT02311842
Title: To Investigate Genetic Factors Associated With the Response to Anti-TNF Therapy in Patients With Early Ankylosing Spondylitis
Brief Title: To Investigate Genetic Factors Associated With the Response to Anti-TNF Therapy in Patients With Early AS
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Gu Jieruo, Professor, Sun Yat-sen University
Other Study IDs: WA1627494
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Ankylosing spondylitits (AS) is a chronic, systemic rheumatic disease primarily affecting spine and sacroiliac joints, which belongs to the group of conditions known as spondyloarthopathies and causes eventual fusion of the spine. Twin study in AS estimated a heritability of over 90%. HLA-B27 is regarded as the earlist and most important gene associated with AS heritability, and over 90% of AS patients carry HLA-B27 gene. HLA-B27 was highly polymorphic, and more than 89 subtypes of B27 gene have been found. Subtypes of HLA-B27 vary between different regions, and so on as the relationship between HLA-B27 subtypes and disease development among different races. Anti-TNF- agents were regarded as one milestone in recent years development on treatment of ankylosing spondylitis, and most patients showed significant improvement after anti-TNF- therapy. Yet part of patients still showed insufficient response. Our previous study suggested AS patients carrying different genotype of SNP in TNF gene had different response to anti-TNF- therapies. But more studies should be carried out to identified more gene polymorphisms associated with treatment response. In this study we designed a prospective, open-label trial to investigate the genetic difference beween AS patients with different response to anti-TNF- therapy. We plan to enroll 50-100 early AS patients which fulfill the 2009 ASAS axial spondyloarthritis classification criteria and have axial symptom for no more than 2 years. The patients must have high disease activity defined as BASDAI 4, and HLA-B27 test must be positive. The patients should be able to receive 24 weeks of etanercept treatment. And patients who have previous other anti-TNF- therapy and any contraindication of anti-TNF- therapy must be excluded. Other medicines should be stable for at least 4 weeks before etanercept treatment begins. For the clinic assessment, patients should fill in the AS questionaires and receive physical examination at each visit. ASAS20 is thought as the primary endpoint. For the genetic polymorphysm detection, we select 10-20 SNP in MHC region associated with AS and 5-10 HLA-B27 subtypes which have been worked over and have definite association with AS. At the first visit 4ml of anticoagulated blood was collected and DNA was extracted. Target SNPs are detected by PCR then direct sequencing. HLA-B27 subtypes are identified using PCRSSP methods. And the relationship between SNPs/HLA-B27 subtypes and different response to anti TNF- therapy is accessed using chi-square statistic process in SPSS software. In this study we plan to investigate the relationship between genetic background and the clinical response to anti-TNF- therapy in AS patients, which has been seldom reported before. Our group have been studying the disease-associated gene of AS for years, and got plenty of data and experience about genetic study of AS.

ELIGIBILITY:
Inclusion Criteria:1.Fulfilled ASAS2009 criterioncriteria; 2.The duration of axial syptoms less than 2 years and in active status before treatment(BASDAI≥4）；3.HLA-B27 positive；4.Completed the Etanercept treatment of 12-24 weeks;5. Completed the clinical data and questionnaire rbefore and after of the treatment; 6. Assigend the ICF. Exclusion Criteria:1. Received other anti-TNF-αagents treatment; 2.Patients with other rheumatic disease which may influent gene test and efficacy, including RA, PsA, OA, SLE, etc. 3.Other possible influence factors , including articular cavity local injections of glucocorticoid prior 4 weeks before TNF alpha antagonists treatment;4. Incomplete data.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients with early AS
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ASAS20 response | 12 weeks

SECONDARY OUTCOMES:
ASAS40/70 response proportion | 12 weeks
ASAS5/6 response proportion | 12 weeks
BASDAI50 response proportion | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jieruo Gu, MD, Principal Investigator — Department of Rheumatology, the Third Affiliated Hospital of Sun Yat-sen University Guangzhou, Guangdong, China
Locations (1):
- Department of Rheumatology, the Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] van der Linden S, Valkenburg H, Cats A. The risk of developing ankylosing spondylitis in HLA-B27 positive individuals: a family and population study. Br J Rheumatol. 1983 Nov;22(4 Suppl 2):18-9. doi: 10.1093/rheumatology/xxii.suppl_2.18. PMID 6606472
- [Background] Brown MA, Kennedy LG, MacGregor AJ, Darke C, Duncan E, Shatford JL, Taylor A, Calin A, Wordsworth P. Susceptibility to ankylosing spondylitis in twins: the role of genes, HLA, and the environment. Arthritis Rheum. 1997 Oct;40(10):1823-8. doi: 10.1002/art.1780401015. PMID 9336417
- [Background] Tam LS, Gu J, Yu D. Pathogenesis of ankylosing spondylitis. Nat Rev Rheumatol. 2010 Jul;6(7):399-405. doi: 10.1038/nrrheum.2010.79. Epub 2010 Jun 1. PMID 20517295
- [Background] Gratacos J, Collado A, Filella X, Sanmarti R, Canete J, Llena J, Molina R, Ballesta A, Munoz-Gomez J. Serum cytokines (IL-6, TNF-alpha, IL-1 beta and IFN-gamma) in ankylosing spondylitis: a close correlation between serum IL-6 and disease activity and severity. Br J Rheumatol. 1994 Oct;33(10):927-31. doi: 10.1093/rheumatology/33.10.927. PMID 7921752
- [Background] Braun J, Bollow M, Neure L, Seipelt E, Seyrekbasan F, Herbst H, Eggens U, Distler A, Sieper J. Use of immunohistologic and in situ hybridization techniques in the examination of sacroiliac joint biopsy specimens from patients with ankylosing spondylitis. Arthritis Rheum. 1995 Apr;38(4):499-505. doi: 10.1002/art.1780380407. PMID 7718003
- [Background] Carter KW, Pluzhnikov A, Timms AE, Miceli-Richard C, Bourgain C, Wordsworth BP, Jean-Pierre H, Cox NJ, Palmer LJ, Breban M, Reveille JD, Brown MA. Combined analysis of three whole genome linkage scans for Ankylosing Spondylitis. Rheumatology (Oxford). 2007 May;46(5):763-71. doi: 10.1093/rheumatology/kel443. Epub 2007 Jan 27. PMID 17259653